CLINICAL TRIAL: NCT06217549
Title: The Effect Of Major Autohemotherapy On Blood Lactate Exchange And Muscle Fatigue In Individuals Exposed To High-Intensity Physical Exercise
Brief Title: Effect of Ozone Therapy on Aerobic Exercise Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Şensu Dinçer, medical doctor, Istanbul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ozone therapy, performance
Record Dates: First submitted 2024-01-09; First posted 2024-01-22 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Ozone Therapy; Exercise Performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy participants (Experimental): healthy, physically active people will be included the study.
  Interventions: Other: ozone therapy

INTERVENTIONS:
Other: ozone therapy — Medical ozone is a mixture of pure ozone gas (0.05-5%) and pure oxygen (99.95-95%). It is produced from pure medical oxygen by medical ozone generators. It is applied to the participants 10 sessions by the intravenous method.

SUMMARY:
The goal of this clinical trial is to investigate the effect of the ozone therapy applied using the major autohemotherapy method on exercise performance in male healthy individuals.

The main question's aims to answer are:

* Is ozone therapy applied with the major autohemotherapy method increase the performance?
* Is ozone therapy applied with the major autohemotherapy method improve the recovery after exercise?
* Participants are asked to continue the same exercise program throughout the study. They were given 10 sessions of ozone therapy over 6 weeks.

Researchers compared the before and after treatment performance and recovery data.

DETAILED DESCRIPTION:
Medical ozone is a mixture of pure ozone gas (0.05-5%) and pure oxygen (99.95-95%). It is produced from pure medical oxygen by medical ozone generators. It is suggested that ozone therapy, which is used to treat a wide variety of diseases and is especially useful in the treatment of tissue ischemia and cardiovascular disorders, creates a mild, temporary and controlled oxidative stress and modulates the antioxidant system and immune system. It was reported that ozone exerted its effects by induction of reactive oxygen species and lipid oxygen products known as ozonides. The therapy modulates the immune system by balancing inflammatory and anti-inflammatory cytokines, increasing antioxidant enzymes and increasing glutathione production. In addition, it increases the production of 2,3-diphosphoglycerate (2,3-DPG) by causing an increase in the rate of red blood cell (RBC) glycolysis, improves red cell rheology, increases the oxidative carboxylation of pyruvate, and activates the hexose monophosphate pathway by stimulating adenosine triphosphate (ATP) production. With a decrease in potential of hydrogen (pH) and a slight increase in 2,3-DPG, the sigmoid curve of oxyhemoglobin shifts to the right due to the Bohr effect. The shift to the right reduces the chemical binding of oxygen to hemoglobin, facilitating oxygen delivery to ischemic tissues. Considering that the most important determinant of exercise performance is tissue oxygenation and that the antioxidant system has a positive effect on fatigue, these data lead to the idea that ozone can improve exercise performance.

There are a few studies in the literature investigating the effect of major ozone treatment on exercise performance. The arguments suggesting that major ozone therapy is effective in exercise performance are based on publications made outside of this subject, which include the mechanism of action of major ozone therapy.

Thus, it was aimed to evaluate the effects of the ozone therapy applied using the major autohemotherapy method on exercise performance with changes in fatigue, exercise duration, blood lactate changes level, anaerobic threshold, and maximal oxygen consumption (VO2max).

ELIGIBILITY:
Inclusion Criteria:

* male
* healthy
* aged between 18-35 years old

Exclusion Criteria:

* suffering from a low back or lower extremity injury or surgical operation in the last one year
* having cardiovascular disease
* having glucose 6 phosphate dehydrogenase enzyme deficiency
* having chronic metabolic disease
* having hyperthyroidism, mental and psychological problems.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2019-08-12 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
VO2max | just before the first ozone therapy session and immediately after the last ozone therapy session
  maximum oxygen consumption, indicator of aerobic capacity, cardiopulmonary exercise tests performed twice for each participant
exercise duration | just before the first ozone therapy session and immediately after the last ozone therapy session
  duration of cardiopulmonary exercise test
Modified Borg Scale | just before the first ozone therapy session and immediately after the last ozone therapy session
  Modified Borg Scale is used to measure the perceived fatigue level. The participants were asked to rate their perceived fatigue on a scale of 1-10. It was expressed as 1 'no fatigue' and 10 'extreme fatigue (exhaustion).
Lactate levels | just before the first ozone therapy session and immediately after the last ozone therapy session
  lactate levels at the end of the each 3-minute grades of each cardiopulmonary exercise tests

CONTACTS AND LOCATIONS:
Locations (1):
- Şensu Dinçer, Istanbul, Turkey (Türkiye)